CLINICAL TRIAL: NCT05521048
Title: Doxycycline Injection of Cutaneous Schwannoma in Neurofibromatosis Type 2
Brief Title: Doxycycline in Cutaneous Schwannoma (NF2)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, D. Bradley Welling, MD, PhD, Professor Harvard Department of Otolaryngology-Head and Neck Surgery, Massachusetts Eye and Ear Infirmary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022P000534
Record Dates: First submitted 2022-08-26; First posted 2022-08-30 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Neurofibromatosis Type 2
Keywords: Cutaneous schwannoma; Doxycycline
MeSH Terms: conditions — Neurofibromatosis 2 | interventions — Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm Open Label (Experimental): Open Label
  Interventions: Drug: Doxycycline Injection [Doxy]

INTERVENTIONS:
Drug: Doxycycline Injection [Doxy] — Injections between 0.1 ml to 4 ml of 10mg/ml doxycycline hyclate will be administered to a maximum of three tumors per patient. The dose administered will be calculated based on tumor size, not to exceed the estimated volume of the tumor or a maximum of 4 ml. Injection of 1% lidocaine may be given pre-doxycycline to reduce injection pain.
  Other Names: Doxycycline Hyclate

SUMMARY:
In this research study the investigators want to learn more about an alternate, local treatment for skin schwannomas. Specifically, local doxycycline intra-tumoral injection will be performed as a potential treatment for NF2-related skin schwannomas, ultimately reducing the risks and costs associated with standard surgical removal of such skin tumors if successful.

DETAILED DESCRIPTION:
Study Design: Interventional Clinical Trial, single-arm, open-label

Estimated Enrollment: Up to 19 participants with NF2-associated cutaneous or subcutaneous schwannomas

Aims: To demonstrate change in peripheral schwannoma size following direct injection into the tumor with doxycycline hyclate.

Nineteen neurofibromatosis type 2-associated peripheral cutaneous or subcutaneous schwannomas between 0.5 cm and 4 cm in greatest diameter will be diagnosed clinically, photographed for documentation of location, and injected with between 0.1 ml to 4 ml of 10mg/ml doxycycline hyclate (Fresenius Kabi, Canton, MA). A maximum of three tumors per patient will be injected. The dose administered will be calculated based on tumor size, not to exceed the estimated volume of the tumor or a maximum of 4 ml. The tumor volume will be estimated by electronic caliper measure of the greatest tumor diameter (D). (V=4/3piR3 where R is the radius (R=D/2) is measured in millimeters and the dose calculated by Vmm3/1000 = injection volume in milliliters). Repeat measures will be made at 6-months and 1-year follow up (+/- 1 month) and documented with electronic calipers and photography. Injection of 1% lidocaine may be given pre-doxycycline to reduce injection pain.

Outcome: The primary outcome will be longitudinal change in tumor maximal diameter measured at 6-months and 1-year compared to baseline defined by a change of 25%. Secondary endpoints include patient reports of paresthesia, pain, skin breakdown or discoloration. Exploratory endpoints will be the change in the sum of maximal diameters.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a confirmed diagnosis of neurofibromatosis 2 by fulfilling National Institute of Health (NIH) criteria or Manchester criteria, or by detection of a causative mutation in the NF2 gene.

   The NIH criteria include presence of:
   * Bilateral vestibular schwannomas, OR
   * First-degree relative with NF2 and EITHER unilateral eighth nerve mass OR
   * Two of the following: neurofibroma, meningioma, glioma, schwannoma, juvenile posterior subcapsular lenticular opacity.

   The Manchester criteria include presence of:
   * Bilateral vestibular schwannomas, OR First-degree relative with NF2 and EITHER unilateral eighth nerve mass OR - Two of the following: neurofibroma, meningioma, glioma, schwannoma, juvenile posterior subcapsular lenticular opacity OR
   * Unilateral vestibular schwannoma AND any two of: neurofibroma, meningioma, glioma, schwannoma, juvenile posterior subcapsular lenticular opacity, OR
   * Multiple meningiomas (two or more) AND unilateral vestibular schwannoma OR
   * Any two of: schwannoma, glioma, neurofibroma, cataract.
2. Patients must have measurable disease, defined as at least one cutaneous/subcutaneous schwannoma with the following qualities:

   * Maximal tumor diameter > 0.5 cm to < 4.0 cm that can be accurately measured by electronic calipers
   * Up to a maximum of 3 tumors/subject may be injected
   * Not located on the face
3. Age ≥ 8 years on day 1 of treatment.
4. Life expectancy of greater than 1 year
5. Lansky/Karnofsky performance status ≥ 60
6. Fully recovered from acute toxic effects of any prior chemotherapy, biological modifiers or radiotherapy
7. Any neurologic deficits must be stable for ≥1 week
8. Patient or parent/legal guardian must be able to provide signed informed consent and assent (as applicable for minors)

Exclusion Criteria:

1. Allergy to doxycycline or tetracycline
2. Tumors located on the face or major motor nerves
3. Patients currently receiving medical anticancer therapies or who have received medical anticancer therapies within 4 weeks of the start of study drug (including chemotherapy and molecular targeted agents), as these may interfere with the study drug
4. Radiation therapy to a study target tumor within 1 year prior to enrollment, or any radiation therapy within 4 weeks prior to enrollment, as these may interfere with our ability to assess response to study drug
5. Prior treatment with any investigational drug within the preceding 4 weeks, as they may interfere with the study drug
6. Unstable or rapidly progressive disease, including patients who require glucocorticoids for symptomatic control of brain or spinal tumors, as this would represent a high risk for inability to comply with the study requirements
7. Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

   * symptomatic congestive heart failure of New York heart Association Class III or IV
   * unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease
   * severely impaired lung function as defined as spirometry and DLCO that is 50% of the normal predicted value and/or O2 saturation that is 90% or less at rest on room air
   * active (acute or chronic) or uncontrolled severe infections liver disease, such as cirrhosis or severe hepatic impairment (Child-Pugh class C)
8. Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods. Adequate contraception (oral contraceptives, contraceptive implants, vaginal ring, or intrauterine devices (IUDs)) must be used at the time of injection but does not need to be carried out past the 1st month of observation.
9. History of significant noncompliance with follow-up that would jeopardize the study evaluation.
10. Patients unwilling to or unable to comply with the study protocol.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2022-09-19 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Tumor Maximal Diameter | 6-months, 1-year
  Longitudinal change in tumor maximal diameter

CONTACTS AND LOCATIONS:
Overall Officials: D. Bradley Welling, MD, PhD, Principal Investigator — Massachusetts Eye and Ear Infirmary
Locations (1):
- Massachusetts Eye and Ear, Boston, Massachusetts, United States

REFERENCES:
- [Background] Ren Y, Chari DA, Vasilijic S, Welling DB, Stankovic KM. New developments in neurofibromatosis type 2 and vestibular schwannoma. Neurooncol Adv. 2020 Nov 16;3(1):vdaa153. doi: 10.1093/noajnl/vdaa153. eCollection 2021 Jan-Dec. PMID 33604573
- [Background] Evans DG. Neurofibromatosis type 2 (NF2): a clinical and molecular review. Orphanet J Rare Dis. 2009 Jun 19;4:16. doi: 10.1186/1750-1172-4-16. PMID 19545378
- [Background] Ostrom QT, Cioffi G, Waite K, Kruchko C, Barnholtz-Sloan JS. CBTRUS Statistical Report: Primary Brain and Other Central Nervous System Tumors Diagnosed in the United States in 2014-2018. Neuro Oncol. 2021 Oct 5;23(12 Suppl 2):iii1-iii105. doi: 10.1093/neuonc/noab200. PMID 34608945
- [Background] Balasubramaniam A, Shannon P, Hodaie M, Laperriere N, Michaels H, Guha A. Glioblastoma multiforme after stereotactic radiotherapy for acoustic neuroma: case report and review of the literature. Neuro Oncol. 2007 Oct;9(4):447-53. doi: 10.1215/15228517-2007-027. Epub 2007 Aug 17. PMID 17704364
- [Background] Coy S, Rashid R, Stemmer-Rachamimov A, Santagata S. Correction to: An update on the CNS manifestations of neurofibromatosis type 2. Acta Neuropathol. 2020 Apr;139(4):667. doi: 10.1007/s00401-019-02044-6. PMID 31432207
- [Background] Petrilli AM, Garcia J, Bott M, Klingeman Plati S, Dinh CT, Bracho OR, Yan D, Zou B, Mittal R, Telischi FF, Liu XZ, Chang LS, Welling DB, Copik AJ, Fernandez-Valle C. Ponatinib promotes a G1 cell-cycle arrest of merlin/NF2-deficient human schwann cells. Oncotarget. 2017 May 9;8(19):31666-31681. doi: 10.18632/oncotarget.15912. PMID 28427224
- [Background] Cosetti MK, Golfinos JG, Roland JT Jr. Quality of Life (QoL) Assessment in Patients with Neurofibromatosis Type 2 (NF2). Otolaryngol Head Neck Surg. 2015 Oct;153(4):599-605. doi: 10.1177/0194599815573002. Epub 2015 Mar 16. PMID 25779467
- [Background] Marchi E, Teixeira LR, Vargas FS. Management of malignancy-associated pleural effusion: current and future treatment strategies. Am J Respir Med. 2003;2(3):261-73. doi: 10.1007/BF03256654. PMID 14720007
- [Background] Godfrey KJ, Kally P, Dunbar KE, Campbell AA, Callahan AB, Lo C, Freund R, Lisman RD. Doxycycline Injection for Sclerotherapy of Lower Eyelid Festoons and Malar Edema: Preliminary Results. Ophthalmic Plast Reconstr Surg. 2019 Sep/Oct;35(5):474-477. doi: 10.1097/IOP.0000000000001332. PMID 30882591
- [Background] Shaye DA, Burks CA, Gadkaree SK, Ncogoza I, Tuyishimire G, Nyabyenda V, Gassore A. Self-compounded Doxycycline Sclerotherapy for the Treatment of Lymphatic Malformations in Low-Resource Settings. World J Surg. 2020 Nov;44(11):3616-3619. doi: 10.1007/s00268-020-05667-z. Epub 2020 Jul 8. PMID 32642795
- [Background] Farnoosh S, Don D, Koempel J, Panossian A, Anselmo D, Stanley P. Efficacy of doxycycline and sodium tetradecyl sulfate sclerotherapy in pediatric head and neck lymphatic malformations. Int J Pediatr Otorhinolaryngol. 2015 Jun;79(6):883-887. doi: 10.1016/j.ijporl.2015.03.024. Epub 2015 Apr 6. PMID 25887132
- [Background] Tang SJ, Sreenarasimhaiah J, Tang L, Rollins N, Purdy PD. Endoscopic injection sclerotherapy with doxycycline for mediastinal and esophageal lymphangiohemangioma. Gastrointest Endosc. 2007 Dec;66(6):1196-200. doi: 10.1016/j.gie.2007.06.023. PMID 18061720
- [Background] Woon JTK, Hoon D, Graydon A, Flint M, Doyle AJ. Aneurysmal bone cyst treated with percutaneous doxycycline: is a single treatment sufficient? Skeletal Radiol. 2019 May;48(5):765-771. doi: 10.1007/s00256-019-03188-y. Epub 2019 Feb 26. PMID 30809704
- [Background] Zhu C, Yan X, Yu A, Wang Y. Doxycycline synergizes with doxorubicin to inhibit the proliferation of castration-resistant prostate cancer cells. Acta Biochim Biophys Sin (Shanghai). 2017 Nov 1;49(11):999-1007. doi: 10.1093/abbs/gmx097. PMID 28985240
- [Background] Alsaadi M, Tezcan G, Garanina EE, Hamza S, McIntyre A, Rizvanov AA, Khaiboullina SF. Doxycycline Attenuates Cancer Cell Growth by Suppressing NLRP3-Mediated Inflammation. Pharmaceuticals (Basel). 2021 Aug 26;14(9):852. doi: 10.3390/ph14090852. PMID 34577552
- [Background] Nicoud IB, Jones CM, Pierce JM, Earl TM, Matrisian LM, Chari RS, Gorden DL. Warm hepatic ischemia-reperfusion promotes growth of colorectal carcinoma micrometastases in mouse liver via matrix metalloproteinase-9 induction. Cancer Res. 2007 Mar 15;67(6):2720-8. doi: 10.1158/0008-5472.CAN-06-3923. PMID 17363593
- [Background] Sagar J, Sales K, Taanman JW, Dijk S, Winslet M. Lowering the apoptotic threshold in colorectal cancer cells by targeting mitochondria. Cancer Cell Int. 2010 Sep 6;10:31. doi: 10.1186/1475-2867-10-31. PMID 20819205
- [Background] Tan Q, Yan X, Song L, Yi H, Li P, Sun G, Yu D, Li L, Zeng Z, Guo Z. Induction of Mitochondrial Dysfunction and Oxidative Damage by Antibiotic Drug Doxycycline Enhances the Responsiveness of Glioblastoma to Chemotherapy. Med Sci Monit. 2017 Aug 26;23:4117-4125. doi: 10.12659/msm.903245. PMID 28842551
- [Background] Reis M, Czupalla CJ, Ziegler N, Devraj K, Zinke J, Seidel S, Heck R, Thom S, Macas J, Bockamp E, Fruttiger M, Taketo MM, Dimmeler S, Plate KH, Liebner S. Endothelial Wnt/beta-catenin signaling inhibits glioma angiogenesis and normalizes tumor blood vessels by inducing PDGF-B expression. J Exp Med. 2012 Aug 27;209(9):1611-27. doi: 10.1084/jem.20111580. Epub 2012 Aug 20. PMID 22908324
- [Background] Zhang L, Xu L, Zhang F, Vlashi E. Doxycycline inhibits the cancer stem cell phenotype and epithelial-to-mesenchymal transition in breast cancer. Cell Cycle. 2017 Apr 18;16(8):737-745. doi: 10.1080/15384101.2016.1241929. Epub 2016 Oct 18. PMID 27753527
- [Background] Sharon D, Cathelin S, Mirali S, Di Trani JM, Yanofsky DJ, Keon KA, Rubinstein JL, Schimmer AD, Ketela T, Chan SM. Inhibition of mitochondrial translation overcomes venetoclax resistance in AML through activation of the integrated stress response. Sci Transl Med. 2019 Oct 30;11(516):eaax2863. doi: 10.1126/scitranslmed.aax2863. PMID 31666400
- [Background] Rok J, Karkoszka M, Rzepka Z, Respondek M, Banach K, Beberok A, Wrzesniok D. Cytotoxic and proapoptotic effect of doxycycline - An in vitro study on the human skin melanoma cells. Toxicol In Vitro. 2020 Jun;65:104790. doi: 10.1016/j.tiv.2020.104790. Epub 2020 Feb 8. PMID 32044399
- [Background] Shen LC, Chen YK, Lin LM, Shaw SY. Anti-invasion and anti-tumor growth effect of doxycycline treatment for human oral squamous-cell carcinoma--in vitro and in vivo studies. Oral Oncol. 2010 Mar;46(3):178-84. doi: 10.1016/j.oraloncology.2009.11.013. Epub 2009 Dec 29. PMID 20036604
- [Background] Hadjimichael AC, Foukas AF, Savvidou OD, Mavrogenis AF, Psyrri AK, Papagelopoulos PJ. The anti-neoplastic effect of doxycycline in osteosarcoma as a metalloproteinase (MMP) inhibitor: a systematic review. Clin Sarcoma Res. 2020 Apr 30;10:7. doi: 10.1186/s13569-020-00128-6. eCollection 2020. PMID 32377334
- [Background] Lee MJ, Hung SH, Huang MC, Tsai T, Chen CT. Doxycycline potentiates antitumor effect of 5-aminolevulinic acid-mediated photodynamic therapy in malignant peripheral nerve sheath tumor cells. PLoS One. 2017 May 30;12(5):e0178493. doi: 10.1371/journal.pone.0178493. eCollection 2017. PMID 28558025
- [Background] Ren Y, Hyakusoku H, Sagers JE, Landegger LD, Welling DB, Stankovic KM. MMP-14 (MT1-MMP) Is a Biomarker of Surgical Outcome and a Potential Mediator of Hearing Loss in Patients With Vestibular Schwannomas. Front Cell Neurosci. 2020 Jul 28;14:191. doi: 10.3389/fncel.2020.00191. eCollection 2020. PMID 32848608
- [Background] Sagers JE, Sahin MI, Moon I, Ahmed SG, Stemmer-Rachamimov A, Brenner GJ, Stankovic KM. NLRP3 inflammasome activation in human vestibular schwannoma: Implications for tumor-induced hearing loss. Hear Res. 2019 Sep 15;381:107770. doi: 10.1016/j.heares.2019.07.007. Epub 2019 Jul 17. PMID 31430634
- [Background] Thalheimer RD, Merker VL, Ly KI, Champlain A, Sawaya J, Askenazi NL, Herr HP, Da JLW, Jordan JT, Muzikansky A, Pearce EM, Sakamoto FH, Blakeley JO, Anderson RR, Plotkin SR; REiNS International Collaboration. Validating Techniques for Measurement of Cutaneous Neurofibromas: Recommendations for Clinical Trials. Neurology. 2021 Aug 17;97(7 Suppl 1):S32-S41. doi: 10.1212/WNL.0000000000012428. Epub 2021 Jul 6. PMID 34230197